CLINICAL TRIAL: NCT01871792
Title: Preventive Effect of the PRetreatment With pItavastatiN on Contrast-Induced Nephropathy in Patients With RenaL Dysfunction UndErgoing Coronary Angiography/Intervention (PRINCIPLE-II Study)
Brief Title: Preventive Effect of Pitavastatin on Contrast-Induced Nephropathy in Patients With Renal Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Gangnam Severance Hospital (Other); Severance Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Myongji Hospital (Other); Bundang CHA Hospital (Other); Inje University (Other); Dankook University (Other); Eulji General Hospital (Other)
Responsible Party: Principal Investigator, Woong Chol Kang, Associate Professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRINCIPLE-II
Record Dates: First submitted 2013-05-25; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Contrast-induced Nephropathy
Keywords: Contrast-induced nephropathy; Prevention; Statin; Pitavastatin
MeSH Terms: interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin (Experimental): Pitavastatin 4 mg/day for 7 days before coronary angiography/intervention
  Interventions: Drug: Pitavastatin
- Placebo (Placebo Comparator): Placebo tablet for 7 days before coronary angiography/intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pitavastatin
  Other Names: Livalo®
  Arms: Pitavastatin
Drug: Placebo — Sugar pill manufactured to mimic Pitavastatin 4 mg tablet
  Arms: Placebo

SUMMARY:
Contrast-induced nephropathy (CIN) is a well-recognized complication of radiographic contrast administration and is associated with increased short- and long-term mortality. Previous strategies including forced diuresis with diuretics or mannitol, intravenous administration of fenoldopam or dobutamine, and postprocedure hemodialysis to prevent CIN have been largely unsuccessful. In addition, the use of N-acetylcysteine to prevent CIN has yielded conflicting outcomes.

A review of a large insurance database and retrospective study have shown that statins therapy is associated with a lower incidence of CIN after percutaneous coronary intervention. The preventive effect of statins on CIN may be attributed to direct pleiotropic effects on the vascular wall such as improvement of endothelial dysfunction, anti-inflammatory or anti-oxidative effect. However, recent randomized trial could not demonstrate the preventive effect of statin on CIN in patients with chronic kidney disease.

Thus, we will investigate the preventive effect of pitavastatin on CIN in patient with renal dysfunction undergoing coronary angiography or intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Need for coronary angiography or intervention in patients with typical symptoms for angina or myocardial infarction, or documented myocardial ischemia at non-invasive studies including ECG, treadmill ECG test, heart spect or coronary CT angiography
* Estimated glomerular filtration rate ≤60 mL/min
* Informed consent

Exclusion Criteria:

* Need for primary percutaneous coronary intervention or emergent intervention in patients with myocardial infarction
* Allergic reaction for contrast agent (Visipaque) or statin
* Contraindication for contrast agent (Visipaque) or statin
* Shock status fron any cause including cardiogenic shock
* Statin use before enrollment (Enrollment after 2 weeks of wash-out period)
* Exposure of contrast agent within 7 days before enrollment
* Pregnancy or Expectation for pregnancy in women of childbearing age
* Heart failure (NYHA class ≥3 or left ventricular ejection fraction < 40%)
* Acute renal injury
* Dialysis therapy
* Mechanical ventilator
* Life expectancy < 6 months
* Non-steroidal anti-inflammatory drug, dopamine, mannitol or N-acetylcysteine, ascorbic acid within 48 hours before and after coronary angiography/intervention
* Severe hepatic dysfunction
* Eisenmenger syndrome or idiopathic pulmonary hypertension
* Renal artery angioplasty within 6 months
* Single functioning kidney
* Kidney transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy | 48 hours
  Contrast-induced nephropathy is defined as either a greater than 25% increase of serum creatinine or an absolute increase in serum creatinine of 0.5 mg/dL after coronary angiography or intervention.

SECONDARY OUTCOMES:
Peak level of serum creatinine | 48 hours
  Peak level of serum creatinine within less than 48 hours after coronary angiography or intervention
serum cystatin-C level | 24 hours
  Absolute level of serum cystatin-C 24 hours after coronary angiography/intervention and Difference level of serum cystatin-C before and after coronary angiography/intervention
serum neutrophil-gelatinase-associated lipocalin(NGAL) level | 4 hours
  Absolute level of serum NGAL level 4 hours after coronary angiography/intervention and difference level before and after coronary angiography/intervention
Length of hospital stay | an expected average of 5 weeks
Clinical events | 1 month
  Composites of death, myocardial infarction, stroke or need for dialysis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Woong Chul Kang, M.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Kang WC, Kim M, Park SM, Kim BK, Lee BK, Kwon HM. Preventive Effect of Pretreatment with Pitavastatin on Contrast-Induced Nephropathy in Patients with Renal Dysfunction Undergoing Coronary Procedure: PRINCIPLE-II Randomized Clinical Trial. J Clin Med. 2020 Nov 17;9(11):3689. doi: 10.3390/jcm9113689. PMID 33213012